CLINICAL TRIAL: NCT06764524
Title: Hairy Cell Leukemia: Harnessing the Full Power of Extracellular Vesicles to Improve Patient Care Management
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EV-ABLE; RC-2024-2790616 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Hairy Cell Leukemia (HCL)
MeSH Terms: conditions — Leukemia, Hairy Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Check whether patients with Hairy Cell Leukemia (HCL) of different status (at diagnosis, in complete remission > 2 years or relapsed requiring therapy) have a 'signature' of altered immunity based on extracellular vesicles (EV)

DETAILED DESCRIPTION:
Extracellular vesicles are small particles detected within plasma and recognized as mediators of intercellular communication thanks to their cargo of proteins, lipids, and nucleic acids. However, the composition of vesicles from Hairy Cell Leukemia patients, which may hold the key to unraveling their involvement and function within tumor microenvironment, is totally unknown. The aim of this study is to characterize these extracellular vesicles in order to identify biology-related and disease-specific biomarkers.

ELIGIBILITY:
Inclusion criteria for patients:

* WHO2022-defined diagnosis of Hairy Cell Leukemia.
* age ≥18 years.
* signed informed consent.

Inclusion criteria for Healthy Donors:

* age ≥18 years.
* Volunteers in general good health, free from any disease or serious illness.
* Signed informed consent.

Exclusion criteria

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed by Hairy Cell Leukemia patients (3 groups: patients at diagnosis (n=10); patients in complete response for >2 years (n=10); relapsed patients meeting treatment indications (n=5)) and by Healthy Donors (n=25) enrolled among volunteers of the no profit organization BolognAIL.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-06-05 (Estimated); Study Completion 2027-12-04 (Estimated)

PRIMARY OUTCOMES:
Extracellular vesicle characterization | 2 years
  Verify whether hairy cell leukemia patients at different status (at diagnosis, in complete remission > 2 years, or relapsed meeting treatment indications) display specific extracellular vesicle-based signatures of immune failure.

SECONDARY OUTCOMES:
Extracellular vesicles' functions and biomarker validation | 2 years
  Elucidate whether immune cells of hairy cell leukemia patients and of healthy donors show specific phenotype. Elucidate whether plasma-derived extracellular vesicles of hairy cell leukemia patients and of healthy donors affect the cross-talk between hairy cells and immune cells. Confirm the biomarkers identified by using bone marrow biopsy of hairy cell leukemia patients, at diagnosis or relapsed meeting treatment indications.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Catani, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy